CLINICAL TRIAL: NCT06911515
Title: Evaluation of Essential Metal Metabolism in Patients With Disorders of Consciousness
Brief Title: Evaluation of Essential Metal Metabolism
Acronym: META-GCA
Status: Active, not recruiting | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, PADUA LUCA, associated professor, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Other Study IDs: 6279
Record Dates: First submitted 2025-03-17; First posted 2025-04-04 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Disturbance of Consciousness; Alteration of Metabolism; Essential Metals
Keywords: patients with disturbance of consciousness; essential metal; metabolism status

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Experimental: Gruop A: Difference in metal concentrations (7 metals) in GCA subjects compared to those in previously acquired sera of healthy controls.
  Interventions: Other: peripheral venous blood samples, these will be performed in order to measure the biological markers in the serum
- Experimental: Group B: Differences and Correlation: Differences in essential metal concentrations at 30 days compared to baseline in GCA patients.
  * Baseline differences in essential metal metabolism in subcategories of patients with impaired consciousness (coma/VS vs MCS, traumatic brain injury vs non-traumatic brain injury).
  * Correlation between clinical scales and essential metal metabolism
  Interventions: Other: peripheral venous blood samples, these will be performed in order to measure the biological markers in the serum

INTERVENTIONS:
Other: peripheral venous blood samples, these will be performed in order to measure the biological markers in the serum — peripheral venous blood samples, these will be performed in order to measure the biological markers in the serum

SUMMARY:
Disturbance of consciousness (DoC) is a state in which consciousness is altered following brain damage and can manifest in several conditions that result from the loss of regulation of the neural function of the two components of consciousness, alertness and awareness.

It is known that the main causes of disorders of consciousness have important effects on the disruption of essential metal homeostasis.

In particular, myocardial infarction and heart failure, ischemic and hemorrhagic stroke and head trauma trigger phenomena of diffuse axonal damage, hypoxia and re-perfusion that profoundly alter the metabolism of cerebral O2 that reacts with essential metals , in Fenton-type reactions whose predominant effect is an extensive production of reactive oxygen species (ROS) and pro-oxidant molecules.

Fe, Cu and zinc (Zn) are essential metals for life: two thirds of the proteins in our body use these metals that play a crucial role as catalysts or structural elements of proteins in various biological processes, such as cellular respiration in mitochondria, the production and maturation of red and white blood cells, the elasticity of connective tissue, the production of myelin and the production of some neurotransmitters. For this reason, the biology of essential metals has a major impact on our health and the disruption of their homeostasis inexorably leads to disease.

These metals are very important for the metabolism of the Central Nervous System (CNS) and Cu, in particular, even in adults, is involved in the production of myelin and in the production of some neurotransmitters of the diffuse modulatory systems . Cu is a cofactor of the enzymes dopamine β-hydroxylase, and monoamine oxidase involved in the balance of catecholamines , and is altered in some disorders of Cu metabolism.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have been in a coma state, documented with a GCS ≤ 8 for at least 24 hours;

  * Presence of a disturbance of consciousness, identified through the Coma Recovery Scale-revised (CRS-r) and classified as coma, vegetative state or minimally conscious state;
  * Latency of the acute event between 15 days and 6 months;
  * Ability of the caregiver/guardian to understand and sign the informed consent.

Exclusion Criteria:

* Age <18 years;

  * Psychiatric or other pathologies;
  * Inflammatory state related to ongoing infections;
  * Refusal or inability to sign the written informed consent to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients of both sexes with DoC being treated at the U.O.C. of High Intensity Neurorehabilitation, Fondazione Policlinico Universitario Gemelli IRCCS of Rome
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2025-03-17 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Blood concetration of essential metal in patients with acquired brain injury | Changes from baseline (T0), after 30 days of treatment (T1)
  Quantification of blood essential metal levels in peripheral venous blood samples in patients with acquired brain injury (Fe, range: Men: 65-178 µg/dL, Women: 50-170 µg/dL; Zn, range: 75- 110 µg/dL; Cu, range: Men: 60-160 µg/dL, Women: 80-155 µg/dL;non-Cp Cu, range: less than 5 µg/dL) compared to healthy patients.

SECONDARY OUTCOMES:
Differences in essential metal blood concentration in subcategories of patients with impaired consciousness | At baseline (T0) and 30 days (T1)
  Baseline differences in essential metal metabolism in subcategories of patients with disturbance of consciousness (coma/VS vs MCS using CRS-r scale range: 0 to 23).
Differences in essential metal blood concentration in subcategories of patients with acquired brain injury (traumatic vs non-traumatic) | At baseline (T0) and 30 days (T1)
  Baseline differences in essential metal blood concentration in subcategories of patients with acquired brain injury ( etiology: traumatic vs non-traumatic).
Correlation between clinical outcome related to autonomy and disability and essential metal blood concentration | At baseline (T0) and 30 days (T1)
  The clinical evaluation will be carried out using the following evaluation scales: Barthel Index (mBI) (range 0 to 100), the Disability Rating Scale (DRS) (range 0 to 29). As regards peripheral venous blood sampling, these will be performed in order to measure the following biological markers on serum: Fe, range men 65 and 178 µg/dL, women 50 and 170 µg/dL; Zn, range 75 -110 µg/dL; Cu, range men 60-160 µg/dL, women: 80-155 µg/dL; Ferr, range men 20-200 ng/mL, women 20-120 ng/mL; Tf, range men: 215-365 mg/dL, women: 250-380 mg/dL; Cp, range 20-50 mg/dL: Non-Cp Cu, range less than 5 µg/dL.
Correlation between clinical outcome related to motor performance and essential metal blood concentration | At baseline (T0) and 30 days (T1)
  The clinical evaluation will be carried out using the following evaluation scales: Motricity Index (range 0 to 100 points). As regards peripheral venous blood sampling, these will be performed in order to measure the following biological markers on serum: Fe, range men 65 and 178 µg/dL, women 50 and 170 µg/dL; Zn, range 75 -110 µg/dL; Cu, range men 60-160 µg/dL, women: 80-155 µg/dL; Ferr, range men 20-200 ng/mL, women 20-120 ng/mL; Tf, range men: 215-365 mg/dL, women: 250-380 mg/dL; Cp, range 20-50 mg/dL: Non-Cp Cu, range less than 5 µg/dL.
Correlation between clinical outcome related to state of consciousness and cognitive level and essential metal blood concentration | At baseline (T0) and 30 days (T1)
  The clinical evaluation will be carried out using the following evaluation scales: Coma Recovery Scale - Journal (CRS-r) (range 0 to 23), the Level of Cognitive Functioning (LCF) (range10 levels) and the Full Outline of UnResponsiveness (FOUR-Score) (range 0 to 16). As regards peripheral venous blood sampling, these will be performed in order to measure the following biological markers on serum: Fe, range men 65 and 178 µg/dL, women 50 and 170 µg/dL; Zn, range 75 -110 µg/dL; Cu, range men 60-160 µg/dL, women: 80-155 µg/dL; Ferr, range men 20-200 ng/mL, women 20-120 ng/mL; Tf, range men: 215-365 mg/dL, women: 250-380 mg/dL; Cp, range 20-50 mg/dL: Non-Cp Cu, range less than 5 µg/dL.

CONTACTS AND LOCATIONS:
Overall Officials: Stefano mr Bonomi, MD,, Study Chair — Fondazione Policlinico Universitario A. Gemelli, IRCCS
Locations (1):
- UOC Neuroriabilitazione ad alta intensità , Policlinico "A. Gemelli", Roma, RM, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Grassi M, Palluzzi F, Tarantino B. SEMgraph: an R package for causal network inference of high-throughput data with structural equation models. Bioinformatics. 2022 Oct 14;38(20):4829-4830. doi: 10.1093/bioinformatics/btac567. PMID 36040154
- [Background] Nicoletti VG, Pajer K, Calcagno D, Pajenda G, Nogradi A. The Role of Metals in the Neuroregenerative Action of BDNF, GDNF, NGF and Other Neurotrophic Factors. Biomolecules. 2022 Jul 22;12(8):1015. doi: 10.3390/biom12081015. PMID 35892326
- [Background] Giacino JT, Kalmar K. Diagnostic and prognostic guidelines for the vegetative and minimally conscious states. Neuropsychol Rehabil. 2005 Jul-Sep;15(3-4):166-74. doi: 10.1080/09602010443000498. PMID 16350959
- [Background] Squitti R, Ventriglia M, Simonelli I, Bonvicini C, Costa A, Perini G, Binetti G, Benussi L, Ghidoni R, Koch G, Borroni B, Albanese A, Sensi SL, Rongioletti M. Copper Imbalance in Alzheimer's Disease: Meta-Analysis of Serum, Plasma, and Brain Specimens, and Replication Study Evaluating ATP7B Gene Variants. Biomolecules. 2021 Jun 29;11(7):960. doi: 10.3390/biom11070960. PMID 34209820
- [Background] Squitti R, Faller P, Hureau C, Granzotto A, White AR, Kepp KP. Copper Imbalance in Alzheimer's Disease and Its Link with the Amyloid Hypothesis: Towards a Combined Clinical, Chemical, and Genetic Etiology. J Alzheimers Dis. 2021;83(1):23-41. doi: 10.3233/JAD-201556. PMID 34219710
- [Background] Cheng L, Cortese D, Monti MM, Wang F, Riganello F, Arcuri F, Di H, Schnakers C. Do Sensory Stimulation Programs Have an Impact on Consciousness Recovery? Front Neurol. 2018 Oct 2;9:826. doi: 10.3389/fneur.2018.00826. eCollection 2018. PMID 30333789
- [Background] Squitti R, Reale G, Tondolo V, Crescenti D, Bellini S, Moci M, Caliandro P, Padua L, Rongioletti M. Imbalance of Essential Metals in Traumatic Brain Injury and Its Possible Link with Disorders of Consciousness. Int J Mol Sci. 2023 Apr 6;24(7):6867. doi: 10.3390/ijms24076867. PMID 37047843
- [Background] Dolce G, Lucca LF, Riganello F, Arcuri F, Quintieri M, Cortese MD, Pignolo L. Advances in the neurorehabilitation of severe disorder of consciousness. Ann Ist Super Sanita. 2014;50(3):234-40. doi: 10.4415/ANN_14_03_06. PMID 25292271
- [Background] von Wild K, Laureys ST, Gerstenbrand F, Dolce G, Onose G. The vegetative state--a syndrome in search of a name. J Med Life. 2012 Feb 22;5(1):3-15. Epub 2012 Mar 5. PMID 22574081
- [Background] Laureys S, Celesia GG, Cohadon F, Lavrijsen J, Leon-Carrion J, Sannita WG, Sazbon L, Schmutzhard E, von Wild KR, Zeman A, Dolce G; European Task Force on Disorders of Consciousness. Unresponsive wakefulness syndrome: a new name for the vegetative state or apallic syndrome. BMC Med. 2010 Nov 1;8:68. doi: 10.1186/1741-7015-8-68. PMID 21040571
- [Background] Davis T, Ings A; National Institute of Health and Care Excellence. Head injury: triage, assessment, investigation and early management of head injury in children, young people and adults (NICE guideline CG 176). Arch Dis Child Educ Pract Ed. 2015 Apr;100(2):97-100. doi: 10.1136/archdischild-2014-306797. Epub 2014 Oct 21. No abstract available. PMID 25335757